CLINICAL TRIAL: NCT03269123
Title: Clinical Trial of a Mechanical Device for the Treatment of Blepharospasm
Brief Title: A Mechanical Device for Blepharospasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: The Dystonia Society of the United Kingdom (Unknown); Globsource UK (Unknown); Statsconsultancy Ltd, Amersham, Buckinghamshire,UK (Unknown)
Responsible Party: Principal Investigator, Alexina Fantato, Principal Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5663
Record Dates: First submitted 2017-08-16; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Blepharospasm
Keywords: Sensory trick; Geste Antagoniste
MeSH Terms: conditions — Blepharospasm

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A device to relieve Blepharospasm (Other): The pressure device known as Pressop1 is the intervention which is attached to the spectacles and worn for 2 weeks prior to retreatment with Botulinum Toxin injections to assess its effectiveness in controlling eyelid spasms.
  Interventions: Device: Pressop 1

INTERVENTIONS:
Device: Pressop 1 — A pressure device attached to the spectacles which mimics a sensory trick (geste Antagoniste)

SUMMARY:
Idiopathic blepharospasm (IB) is a rare but well characterised adult onset focal dystonia that may cause severe visual disability. The most effective treatment is with periodic injections of botulinum toxin into the pre-tarsal and / or pre-septal orbicularis oculi muscles bilaterally. However, even with treatment, practical visual function often remains compromised.

A subset of IB sufferers find that eye opening improves with focal unilateral digital pressure usually on a specific point on the temple. The Investigators have developed a spectacle mounted spring-loaded prosthesis (the "Pressop" device) to apply continuous individually localised focal pressure on the temple to mimic the effect of finger pressure.

The Investigators recommended a trial of this simple safe device in those IB patients who report improvement in eye opening with focal digital temple pressure.

DETAILED DESCRIPTION:
Idiopathic blepharospasm is a rare chronic neuro-ophthalmic disorder that causes substantial visual handicap & compromises quality of life. It affects adults, women more than men, usually beginning in the 5th or 6th decade and consists of repeated forceful bilateral spasms of eye closure with photophobia and ocular surface discomfort. In up to a third of cases there are synchronous mid and / or lower facial spasms and the spectrum of disorder extends to cranial dystonia involving jaw & neck muscle spasms (e.g. antecollis or retrocollis). Practical visual function is variably affected but most patients will have to stop driving, many cannot work, manage the house or even leave the house unaccompanied. Leisure activities such as reading & watching television are compromised or impossible, and secondary mood dysphoria and depression are common.

In some cases, patients have discovered that applying focal finger pressure, usually to the temple, relieves or even abolishes the spasms for the duration of the application. It is, however, difficult for the patient to sustain the finger pressure and impossible to apply it during activities when eyesight is important e.g. driving, typing or other bimanual tasks. The phenomenon can be regarded as the equivalent of the sensory trick (ST or geste antagonistique) seen in some cases of spasmodic torticollis whereby finger tip pressure on the chin prevents or reduces the muscle spasms in the neck and allows the head to be held straight.

In this study, the Investigators explored the hypothesis that the benefit of the finger-tip pressure sensory trick could be replicated by a spring-loaded, spectacle mounted device applying focal pressure to the temple. Following preliminary design trials, the investigators commissioned a manufacturer to develop a light easily handled pressure device that could be fixed to the frame of most spectacles. The "Pressop" device fulfils these criteria and was adopted for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient with Blepharospasm of sufficient severity to necessitate repeated Botulinum injections can be included in the study.
* It is not essential for participants to be spectacle wearers (having a refractive error) as prescription free (zero power) spectacles can be provided for the purposes of being able to trial the device .
* The participants may or may not be currently having Botulinum Toxin injections. Some of these patients will be known to use the "Geste Antagoniste" phenomenon. Patients who may not know of this potential therapeutic effect will also be invited to trial the device.

Exclusion Criteria:

* Inability to wear spectacles due to any reason (as the device has to be mounted on the spectacle frame).
* Patients who have spasms and twitches of the eyes caused by a different pathology e.g. Hemi facial Spasm, Parkinson's disease will also be excluded from this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03-02 (Actual); Primary Completion 2011-08-08 (Actual); Study Completion 2011-08-08 (Actual)

PRIMARY OUTCOMES:
The study's objective and subjective responses for the use of the device is measured with the CDQ-24 questionnaire and a questionnaire specific to the the device | 2-3 week trial period
  Outcome measures will be taken from the CDQ-24 assessment carried out before and after using the pressure device demonstrating improved quality of life.The questionnaire specific to the device addresses issues like wearing time, discomfort, suggestions and feedback .

SECONDARY OUTCOMES:
The proportion of patients demonstrating the "Geste Antagoniste" phenomenon. | 2-3 week trial period
  This proportion will be presented, along with its 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: John S Elston, MD FRCS OPTH, Study Director — Oxford University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
The study findings will be published in the appropriate medical journal